CLINICAL TRIAL: NCT03715894
Title: Edwards SAPIEN 3 PPI Registry - A Retrospective Survey and Prospective Identification of Procedure Related Variables Associated With Permanent Pacemaker Implantation in Patients Receiving an Edwards SAPIEN 3 Valve
Brief Title: Prospective Arm of Conduct - Edwards SAPIEN3 PPI Registry
Acronym: Conduct-pro
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: Conduct prospective
Record Dates: First submitted 2018-10-02; First posted 2018-10-23 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Aortic Valve Stenosis; AV Block; Bundle-Branch Block
Keywords: Transcatheter aortic valve implantation; Pacemaker; Aortic valve calcification; PPI
MeSH Terms: conditions — Aortic Valve Stenosis; Atrioventricular Block; Bundle-Branch Block; Aortic Valve, Calcification of | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with aortic stenosis: Patients receiving Edwards SAPIEN 3 aortic transcatheter valve Implantation, who are with a high risk for PPI
  Interventions: Procedure: transcatheter valve implantation

INTERVENTIONS:
Procedure: transcatheter valve implantation — aortic transcatheter valve implantation using Edwards SAPIEN 3 valve

SUMMARY:
There are procedure related risk factors for permanent pacemaker implantation (PPI) that can be identified and assessed in a prospective cohort of 300 patients at high risk for PPI

Prospective, multicenter, European registry in patients at high risk for PPI undergoing TAVI with the Edwards SAPIEN 3 valve. Additional assessment of calcification using a CT data core lab. Statistical analysis of the dataset obtained with respect to the objectives of the registry.

DETAILED DESCRIPTION:
Permanent pacemaker implantation is a widely recognized clinical event associated with TAVI becoming evident within a few days after the procedure.

While a number of registries have documented the rates of PPI with different valves, much less evidence has been provided for

1. patient based characteristics (e.g. RBBB etc.) affecting the likelihood of PPI and for
2. procedural variables (e.g. implantation hieght, valve size etc.) that should be considered to perform as safe and minimal invasive procedure as possible.

Prior Research To date there are 8 published reports on pacemaker rates and predictors associated with the use of the Edwards SAPIEN 3 THV.

These studies suggest that the need for pacemaker implantation in single centers ranges between 14.4 and 20.4% based on patient numbers between 131 and 335 patients.

These analyses resulted in the identification of pre-existing conduction disturbance, aortic valve calcification, heavily calcified LVOT, RBBB, persistent complete heart blocks, prolonged QRS duration or short membranous septum as patient related factors associated with PPI during Edwards SAPIEN 3 THV TAVI. Similarly, procedural variables such as implantation height /oversizing as procedure related variables are associated with PPI after TAVI.

The literature regarding procedure related variables associated with permanent pacemaker implantation in patients receiving an Edwards SAPIEN 3 valve shows multivariable analyses with slightly different views to the requested procedural variables.

Tarantini et al. suggest a higher valve implantation (ventricular ratio >60/40 at qualitative assessment or depth <8mm at qualitative assessment). A similar outcome was reported by De Torres-Alba et al.. Due to the longer stent of the SAPIEN 3 they suggest an even higher implantation, intending a shorter extension of the stent into the LVOT by increasing the percentage of the stent in the aorta to >70%. Schwerg et al. compare the PPI rate in "low implantation" with "high implantation" independently from the patients pre-existing conduction disturbances, and suggest to minimize the risk of PPI by choosing a higher implantation technique with the central marker 2 mm or more over the annular plane.

Furthermore Mauri et al. encourage to choose a implantation height of <25.5% (Implantation height was expressed as the percentage of the ventricular part of the stent frame in relation to the overall stent frame length).

Another procedural factor is found to be aortic annulus oversizing ratios which are known to prevent paravalvular leakage. Leber et al. show the rate of post-procedural permanent pacemakers tended to be lower in patients with <15% oversizing compared to those with >25% oversizing for Edwards Sapien XT. Using SAPIEN 3 valves Husser et al. show a higher PPI rate in patients with out of range oversizing.

Gonska et al. conclude that neither implantation height nor oversizing has an effect on PPI rate.

On the other hand the need for pre-dilatation by balloon valvuloplasty and post-implant dilatation have not been identified as potential contributing factors for PPI as it is believed the impact of the dilatation on the conduction tissue is transient and short lived.

Nevertheless, pre- and post-dilatation should be further considered and analysed.

Hypothetically, also the following procedural parameters, which have not been investigated in detail so far, could be risks for PPIs: Stiff guidewire use or a no touch policy and should be considered in this research.

Limitations of prior research Current evidence though is limited by patient numbers versus event rates (with a max. of 62 PPI considered in any of the available datasets) resulting in a limited power in multivariable analyses, the single center design of these ventures, the lack of a consistent definition of variables potentially associated with PPI and the unexplained differences in the number and type of variables identified.

Aims This registry aims to assess procedural variables and to verify risk factors in a prospective multicenter registry.

To identify predictors of PPI patients with a high risk for PPI will be preferably included to increase the power compared to pre-existing database analyses from single centres. The target is to identify general procedural predictors and to verify risk factors of PPI post TAVI with the Edwards SAPIEN 3 valve which when identified and avoided will reduce the need of PPI in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing transfemoral SAPIEN 3 implantation because of aortic stenosis,
* at least 1 of the identified risk factors from the retrospective part to ensure a minimum risk of 33% for PPI (presumed: pre-existing conduction disturbance, aortic valve calcification, heavily calcified LVOT, RBBB, persistent complete heart blocks, QRS duration or short membranous septum,to be confirmed);

Exclusion Criteria:

* exclusion of patients with prior pacemaker,
* with indications for pacemaker implantation prior to TAVI
* valve in valve implantation or
* without informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing transfemoral transcatheter valve implantation with the SAPIEN 3 valve with at least one identified risk factor for PPI
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Occurence of permanent pacemaker implantation after TAVI in high risk patients | 1 year
  Need for permanent pacemaker implantation after TAVI in high risk patients.

SECONDARY OUTCOMES:
Implantation depth | up to 30 days after intervention
  Measurement in peri-interventional aortic angiograms. Mean implantation depth (% ventricular part of the stent frame)
Valve sizing | up to 30 days after intervention
  Measurement of aorta in pre-operative contrast multislice computed tomographic Images, compared to the implanted valve sizing. Percentage of oversizing will be calculated using the formula (nominal prosthesis area/multislice computed tomographic area - 1) x 100
Dilatation | 1 year
  Ratio in patients, who get a dilatation before or at intervention as well as thereafter (discharge, FU)
Expiration data | 2 years
  cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Geisler, Prof., Principal Investigator — University Clinic Tübingen, Tübingen, Germany - Department of Internal Medicine III
Locations (5):
- Germany (3):
  - University Clinic Tübingen, Department of Internal Medicine III, Tübingen, Baden-Wurttemberg
  - University Clinic Ulm, Department of Internal Medicine II, Ulm, Baden-Wurttemberg
  - Herz- und Diabeteszentrum, Bad Oeynhausen, North Rhine-Westphalia
- Academisch Medisch Centrum (AMC), Amsterdam, Netherlands
- Dept of Cardiology, Linköping University Hospital,, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No
no IPD will be made available

REFERENCES:
- [Background] Bob-Manuel T, Nanda A, Latham S, Pour-Ghaz I, Skelton WP 4th, Khouzam RN. Permanent pacemaker insertion in patients with conduction abnormalities post transcatheter aortic valve replacement: a review and proposed guidelines. Ann Transl Med. 2018 Jan;6(1):11. doi: 10.21037/atm.2017.10.21. PMID 29404357
- [Background] De Torres-Alba F, Kaleschke G, Diller GP, Vormbrock J, Orwat S, Radke R, Reinke F, Fischer D, Reinecke H, Baumgartner H. Changes in the Pacemaker Rate After Transition From Edwards SAPIEN XT to SAPIEN 3 Transcatheter Aortic Valve Implantation: The Critical Role of Valve Implantation Height. JACC Cardiovasc Interv. 2016 Apr 25;9(8):805-813. doi: 10.1016/j.jcin.2015.12.023. Epub 2016 Mar 23. PMID 27017367
- [Background] Maeno Y, Abramowitz Y, Kawamori H, Kazuno Y, Kubo S, Takahashi N, Mangat G, Okuyama K, Kashif M, Chakravarty T, Nakamura M, Cheng W, Friedman J, Berman D, Makkar RR, Jilaihawi H. A Highly Predictive Risk Model for Pacemaker Implantation After TAVR. JACC Cardiovasc Imaging. 2017 Oct;10(10 Pt A):1139-1147. doi: 10.1016/j.jcmg.2016.11.020. Epub 2017 Apr 12. PMID 28412434
- [Background] Tarantini G, Mojoli M, Purita P, Napodano M, D'Onofrio A, Frigo A, Covolo E, Facchin M, Isabella G, Gerosa G, Iliceto S. Unravelling the (arte)fact of increased pacemaker rate with the Edwards SAPIEN 3 valve. EuroIntervention. 2015 Jul;11(3):343-50. doi: 10.4244/EIJY14M11_06. PMID 25405801
- [Background] Mauri V, Reimann A, Stern D, Scherner M, Kuhn E, Rudolph V, Rosenkranz S, Eghbalzadeh K, Friedrichs K, Wahlers T, Baldus S, Madershahian N, Rudolph TK. Predictors of Permanent Pacemaker Implantation After Transcatheter Aortic Valve Replacement With the SAPIEN 3. JACC Cardiovasc Interv. 2016 Nov 14;9(21):2200-2209. doi: 10.1016/j.jcin.2016.08.034. PMID 27832845
- [Background] Gonska B, Seeger J, Kessler M, von Keil A, Rottbauer W, Wohrle J. Predictors for permanent pacemaker implantation in patients undergoing transfemoral aortic valve implantation with the Edwards Sapien 3 valve. Clin Res Cardiol. 2017 Aug;106(8):590-597. doi: 10.1007/s00392-017-1093-2. Epub 2017 Mar 10. PMID 28283746
- [Background] Husser O, Pellegrini C, Kessler T, Burgdorf C, Thaller H, Mayr NP, Kasel AM, Kastrati A, Schunkert H, Hengstenberg C. Predictors of Permanent Pacemaker Implantations and New-Onset Conduction Abnormalities With the SAPIEN 3 Balloon-Expandable Transcatheter Heart Valve. JACC Cardiovasc Interv. 2016 Feb 8;9(3):244-254. doi: 10.1016/j.jcin.2015.09.036. PMID 26847116
- [Background] Schwerg M, Fulde F, Dreger H, Poller WC, Stangl K, Laule M. Optimized Implantation Height of the Edwards SAPIEN 3 Valve to Minimize Pacemaker Implantation After TAVI. J Interv Cardiol. 2016 Aug;29(4):370-4. doi: 10.1111/joic.12302. Epub 2016 May 31. PMID 27240558
- [Background] Fujita B, Kutting M, Seiffert M, Scholtz S, Egron S, Prashovikj E, Borgermann J, Schafer T, Scholtz W, Preuss R, Gummert J, Steinseifer U, Ensminger SM. Calcium distribution patterns of the aortic valve as a risk factor for the need of permanent pacemaker implantation after transcatheter aortic valve implantation. Eur Heart J Cardiovasc Imaging. 2016 Dec;17(12):1385-1393. doi: 10.1093/ehjci/jev343. Epub 2016 Jan 12. PMID 26758411